CLINICAL TRIAL: NCT04139837
Title: Frailty in Daily Practice: Screening, Consultation and Education Activities
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jean Woo, Professor, Chinese University of Hong Kong
Other Study IDs: 2019.475
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Health screening, community health talks or activities on frailty — Screening for frailty using the FRAIL scale to categorize participant's status as robust, prefrail and frail. A series of community health talks or activities on frailty will be provided to each category of participants for the prevention or management of frailty.

SUMMARY:
The present study is designed to to estimate the prevalence of frailty and pre-frailty and their associated factors in community-dwelling populations aged 50 years and above in Hong Kong, and to explore the views of participants taking part in a community health talks or activities on frailty about what the participants felt or had gained from participating, concerns, and suggestions for change or improvement.

A survey of 15000 people aged 50 years or older identified in community facilities will be conducted. The participants will be invited to their affiliated centres for a brief screening using the FRAIL scale and assessment. A series of community health talks or activities on frailty will be offered to the participants based on the frailty status.Questionnaire and screening tools will be administered by trained researchers.

DETAILED DESCRIPTION:
A 30-month community survey will be conducted, and the survey will be divided into three phases, namely study preparation and subject recruitment (6 months), data collection (18 months), and data entry and analysis (6 months).

A survey of 15000 people aged 50 years or older identified in community facilities (e.g., neighbourhood elderly centre, social centre for the elderly) will be conducted. The participants will be invited to their affiliated centres for a brief screening using the FRAIL scale and assessment. A series of community health talks or activities on frailty will be offered to the participants based on the frailty status. Questionnaire and screening tools will be administered by trained researchers.

The primary outcome will be the prevalence of frailty and pre-frailty. Secondary outcomes will cover physical performance measures including hand-grip strength and 5-chair stand test. Anthropometric and demographic data will also be collected using standardized methods and questionnaires respectively.

Views of participants taking part in a community health talks or activities on frailty about what the participants felt or had gained from participating, concerns, and suggestions for change or improvement will be explored by client satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* People aged 50 years or older
* Chinese origin
* Normally reside in Hong Kong
* Could speak and understand Chinese
* Willing to follow the study procedures

Exclusion Criteria:

-Live in a residential aged care facility

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People aged 50 years or older will be identified in community facilities (e.g., neighbourhood elderly centre, social centre for the elderly).
Sampling Method: Non-Probability Sample
Enrollment: 5951 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Frailty status | 1 day (Once only at screening)
  Frailty status (i.e. robust, prefrail or frail) measured using the frailty scale (FRAIL) in which unabbreviated scale name is unavailable for this scale. Frailty scores from 0 to 5 (i.e., 1 point for each component; 0 = best to 5 = worst) and represent robust (0), pre-frail (1-2), and frail (3-5) health status.

SECONDARY OUTCOMES:
Handgrip strength | 1 day (Once only at screening)
  Handgrip strength measured using a dynamometer
5 chair stands | 1 day (Once only at screening)
  Muscle endurance in the lower extremities - Participant will be required to rise from a chair a total of 5 times, as quickly as they could, with arms across their chest. The amount of time required to complete all 5 repetitions will be recorded.

OTHER OUTCOMES:
Weight | 1 day (Once only at screening)
  Weight in kilogram measured using standardized method
Height | 1 day (Once only at screening)
  Height in centimeter measured using standardized method
Waist circumference | 1 day (Once only at screening)
  Waist circumference in centimeter measured using standardized method
Systolic blood pressure | 1 day (Once only at screening)
  Systolic blood pressure in mmHg measured using standardized method
Diastolic blood pressure | 1 day (Once only at screening)
  Diastolic blood pressure in mmHg measured using standardized method

CONTACTS AND LOCATIONS:
Overall Officials: Jean Woo, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China